CLINICAL TRIAL: NCT03793452
Title: Effect of Pulmonary Rehabilitation on Fear of Falling in COPD Patients
Acronym: PARACHUTE
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: PARACHUTE (29BRC18.0246)
Record Dates: First submitted 2019-01-02; First posted 2019-01-04 (Actual); Last update posted 2020-07-16 (Actual); Status verified 2020-07

CONDITIONS: Copd
Keywords: COPD, pulmonary rehabilitation, fear of falling, evaluation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to measure the impact of pulmonary rehabilitation program on fear of falling in COPD patients

ELIGIBILITY:
Inclusion Criteria:

* COPD patients

Exclusion Criteria:

* post surgical rehabilitation
* neurologic or orthopedic disorders limiting walking
* imbalance disorders
* inability to answer to the questionnaire
* refusal to participate.
* inability to perform the pulmonary rehabilitation program.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: COPD patients admitted for pulmonary rehabilitation program in pulmonary rehabilitation unit of CH des Pays de Morlaix
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2019-01-18 (Actual); Primary Completion 2019-12-18 (Actual); Study Completion 2019-12-18 (Actual)

PRIMARY OUTCOMES:
measure of fear of falling after a pulmonary rehabilitation | 4 weeks
  measure of fear of falling (FES-I) before and after a pulmonary rehabilitation program

CONTACTS AND LOCATIONS:
Overall Officials: Marc Beaumont, PhD, Principal Investigator — CH DES PAYS DE MORLAIX
Locations (1):
- CH Pays de Morlaix, Morlaix, France

REFERENCES:
- [Derived] Berriet AC, Beaumont M, Peran L, Le Ber C, Couturaud F. Effects of pulmonary rehabilitation on fear of falling in Chronic Obstructive Pulmonary Disease (COPD) patients: An observational study. Respir Med Res. 2022 Nov;82:100932. doi: 10.1016/j.resmer.2022.100932. Epub 2022 Jun 12. PMID 35878569